CLINICAL TRIAL: NCT06535542
Title: A Randomized Trial of Integrating Whole Genome Sequencing and Digital Twins Into the Management of Hypercholesterolemia in Emiratis
Brief Title: Integrating Whole Genome Sequencing and Digital Twins Into the Management of Hypercholesterolemia in Emiratis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abu Dhabi Health Services Company (Other Government)
Collaborators: Predictiv Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: WGS_DT_2023; DOH/CVDC/2023/926 (Other Grant/Funding Number: Abu Dhabi Department of Health (DOH))
Record Dates: First submitted 2024-06-28; First posted 2024-08-02 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Hypercholesterolemia, Autosomal Dominant; Hypercholesterolemia, Autosomal Recessive; Familial Combined Hypercholesterolemia
Keywords: LDH; Familial Hypercholesterolemia; Whole Genome Sequencing; Digital Twins; Management of Hypercholesterolemia; Emirati; Randomized Controlled Trial; Sanger Sequencing; Predictiv Care; Genomic Medicine; Precision Medicine; Pharmacogenomics
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hyperlipoproteinemia Type III | interventions — Whole Genome Sequencing

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial of whole-genome sequencing.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigative site personnel will obtain the subject's identification number and study treatment assignment from the randomizer. Participants and all personnel directly involved in the study conduct will be blinded to the arm assignment until 2-3 months after enrollment when the whole-genome sequencing (WGS) report is generated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WGS + Digital Twin Group (Experimental): 20 participants who are randomized to have whole-genome sequencing performed on their sample and given access to Predictiv™ Digital Twin. These participants will meet with a genetic counselor for results disclosure and training to access the Predictiv™ Digital Twin platform.
  Interventions: Genetic: Whole Genome Sequencing
- Standard of Care Group (No Intervention): 20 participants who are randomized to not have whole-genome sequencing performed on their sample. These participants will have standard-of-care familial hypercholesterolemia (FH) evaluation using medical history and family history only. They will not receive genetic results or Predictiv™ Digital Twin results as part of this study.

INTERVENTIONS:
Genetic: Whole Genome Sequencing — Participants in this arm will have their blood sample analyzed by whole-genome sequencing (WGS) and will be given access to Predictiv™ Deoxyribonucleic acid (DNA)-based digital twin platform, a web-based interactive application with WGS results. The platform will include positive monogenic and polygenic Familial Hypercholesterolemia results and pharmacogenomics results on statins and clopidogrel. A report of positive monogenic variants will be included in their medical record. This may also include genes on the American College of Medical Genetics and Genomics (ACMG) secondary findings (SF) version 3.2 list if the participant consents to receive these incidental findings. The report will only include pathogenic, likely pathogenic, and variant of uncertain significance (VUS) results.
  Arms: WGS + Digital Twin Group

SUMMARY:
This pilot study investigates integrating whole genome sequencing and digital twin technology for managing hypercholesterolemia in Abu Dhabi clinics. It aims to establish protocols for larger future studies and incorporate genomic insights into routine medical care.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is the leading cause of death in the Middle East, with hypercholesterolemia being a significant contributor. Genetic mechanisms of hypercholesterolemia in this region are not well understood. Autosomal dominant hypercholesterolemia is a major factor, yet only ~7% of Emiratis with familial hypercholesterolemia (FH) have these mutations. In 2013, Talmud et al. identified common variants through genome-wide association studies (GWAS) that suggest a polygenic cause for hypercholesterolemia in mutation-negative FH patients. A polygenic risk score based on 12 SNPs was validated in White European populations and is used in the UK's NHS diagnostic pipeline. Distinguishing polygenic hypercholesterolemia from FH without genetic testing is challenging. These patients exhibit familial moderate hypercholesterolemia and early coronary heart disease, with elevated LDL-C, normal triglycerides, and no tendon xanthoma. Their cardiovascular risk is similar to monogenic FH with age.

Statins, though commonly prescribed for ASCVD prevention, can cause musculoskeletal symptoms leading to poor adherence, discontinuation, elevated cholesterol, and increased cardiovascular risk. Many patients fail to achieve target LDL-C levels due to suboptimal dosing. Certain gene variants increase the risk of statin side effects.

This study seeks to integrate whole genome sequencing (WGS) technology in a clinical setting through an innovative digital twin platform. This platform allows clinicians to assess monogenic and polygenic risks in real-time and make informed statin prescribing and management decisions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 2 or more LDL-C levels greater than 190 mg/dL or 5.0 mmol/L in the past 12 months
* Undiagnosed patients meeting Possible, Probable or Definitive FH criteria according to Dutch Lipid Clinic Network (DLCN) criteria (Eur Heart J. 2011 Jul;32(14):1769-818. doi: 10.1093/eurheartj/ehr158. Epub 2011 Jun 28.)
* Patients who have not been on anti-lipidemic medication in the past 3 months
* Ages 18-55
* Emirati national
* All patients must be fluent in English or Arabic

Exclusion Criteria:

* - Patients who do not meet the above criteria
* Patients with a previous diagnosis of FH
* Patients with a progressive debilitating illness
* Patient with untreated hypothyroidism, history of proteinuria, obstructive liver disease, chronic renal failure, human immunodeficiency virus infection, or on immunosuppressant or steroid or psychiatric medications
* Patients with untreated clinical anxiety or depression (as measured by a Hospital Anxiety and Depression Scale (HADS) score of ≥ 16 on the depression subscale)
* Patients who are pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic capabilities | From consent date until first documented report, up to 6 months
  Diagnostic yield of standard-of-care (based on medical and family history) versus whole genome sequencing (WGS) for identifying monogenic and polygenic familial hypercholesterolemia.

SECONDARY OUTCOMES:
Prognostic capabilities of standard-of-care | Baseline to End of Study, up to 12 months
  Prognostic capabilities of standard-of-care (based on medical and family history) versus whole genome sequencing for predicting outcomes and management in monogenic and polygenic familial hypercholesterolemia.
Resources Implementation for WGS in a clinical setting | Baseline to End of Study, up to 12 months
  Assessed by documenting resources necessary for each phase, including execution of WGS, reporting of results, and overall evaluation,
Participant characteristics | Baseline
  Age, sociodemographic, personal and family history
Change in Perceived Utility | Baseline, post-disclosure of results (approximately 2-3 months after enrollment), 6 months post-enrollment
  Assessed using novel participant surveys via questions including: attitudes towards DNA testing and results, understanding of results, change in expectations, confidence, concerns.
Changes in Health Care Utilization | Baseline to End of Study, up to 12 months
  Assessed by reviewing medical records comparing number of services and procedures received related to the diagnosis.
Clinician Attitudes About WGS | Baseline
  A self-built survey was created to assess physicians' perspective and attitude toward WGS

CONTACTS AND LOCATIONS:
Overall Officials: Abdulmajeed BS Alzubaidi, MD, Principal Investigator — Abu Dhabi Health Services Co. -SEHA; Erik J Koornneef, PHD, Study Director — Abu Dhabi Health Services Co. -SEHA; Mhy-Lanie Adduru, MD, Study Director — Predictiv Care, Inc.; Salah Eldin HM Hu, MD, Study Chair — Abu Dhabi Health Services Co. -SEHA
Locations (1):
- Abu Dhabi Health Research Center, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Data requests can be submitted 9 months after article publication, and the data will be made accessible for up to 12 months. Extensions will be considered on a case-by-case basis.
Supporting Information: SAP, CSR
Time Frame: 9-12 months
Access Criteria: Qualified researchers engaged in independent scientific research can request access to trial IPD, which will be provided following the review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact mhy-lanie@predictivcare.com.

REFERENCES:
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Wang J, Dron JS, Ban MR, Robinson JF, McIntyre AD, Alazzam M, Zhao PJ, Dilliott AA, Cao H, Huff MW, Rhainds D, Low-Kam C, Dube MP, Lettre G, Tardif JC, Hegele RA. Polygenic Versus Monogenic Causes of Hypercholesterolemia Ascertained Clinically. Arterioscler Thromb Vasc Biol. 2016 Dec;36(12):2439-2445. doi: 10.1161/ATVBAHA.116.308027. Epub 2016 Oct 20. PMID 27765764
- [Background] Futema M, Bourbon M, Williams M, Humphries SE. Clinical utility of the polygenic LDL-C SNP score in familial hypercholesterolemia. Atherosclerosis. 2018 Oct;277:457-463. doi: 10.1016/j.atherosclerosis.2018.06.006. PMID 30270085
- [Background] Talmud PJ, Shah S, Whittall R, Futema M, Howard P, Cooper JA, Harrison SC, Li K, Drenos F, Karpe F, Neil HA, Descamps OS, Langenberg C, Lench N, Kivimaki M, Whittaker J, Hingorani AD, Kumari M, Humphries SE. Use of low-density lipoprotein cholesterol gene score to distinguish patients with polygenic and monogenic familial hypercholesterolaemia: a case-control study. Lancet. 2013 Apr 13;381(9874):1293-301. doi: 10.1016/S0140-6736(12)62127-8. Epub 2013 Feb 22. PMID 23433573
- [Background] Rimbert A, Daggag H, Lansberg P, Buckley A, Viel M, Kanninga R, Johansson L, Dullaart RPF, Sinke R, Al Tikriti A, Kuivenhoven JA, Barakat MT. Low Detection Rates of Genetic FH in Cohort of Patients With Severe Hypercholesterolemia in the United Arabic Emirates. Front Genet. 2022 Jan 3;12:809256. doi: 10.3389/fgene.2021.809256. eCollection 2021. PMID 35047021
- [Background] Bamimore MA, Zaid A, Banerjee Y, Al-Sarraf A, Abifadel M, Seidah NG, Al-Waili K, Al-Rasadi K, Awan Z. Familial hypercholesterolemia mutations in the Middle Eastern and North African region: a need for a national registry. J Clin Lipidol. 2015 Mar-Apr;9(2):187-94. doi: 10.1016/j.jacl.2014.11.008. Epub 2014 Nov 29. PMID 25911074
- See also: The Human Genome Project Completion: Frequently Asked Questions. — http://www.genome.gov/11006943
- See also: Catalog of Published Genome-Wide Association Studies. — http://www.genome.gov/gwastudies/
- See also: Checklists for improving rigour in qualitative research: a case of the tail wagging the dog? — http://doi.org/10.1136/bmj.322.7294.1115
- See also: The West Midland Familial Hypercholesterolaemia (FH) screening programme: Evaluating the utility of the 12 SNP polygenic risk score (PRS) across ethnic groupings — https://doi.org/10.1016/j.athplu.2021.07.012